CLINICAL TRIAL: NCT03511508
Title: Efficacy of a Midwife-coordinated, Individualized, and Specialized Maternity Care Intervention (ChroPreg) in Addition to Standard Care in Pregnant Women With Chronic Disease: a Parallel Randomized Controlled Trial
Brief Title: Pregnancy and Chronic Disease: The Effect of a Midwife-coordinated Maternity Care Intervention
Acronym: ChroPreg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Kristine Hegaard, Midwife, ph.d. Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChroPreg
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Chronic Diseases in Pregnancy
Keywords: pregnancy; maternity Care; complex intervention; interdisiplinary team; chronic disease; interdisciplinary; midwifery
MeSH Terms: conditions — Chronic Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Intervention Group and Control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChroPreg (Active Comparator): The participants in the intervention Group receive the midwife-coordinated, individualized and specialized intervention plus standard care
  Interventions: Behavioral: ChroPreg + standard care
- Standard care alone (No Intervention): Participants in the control group receive the standard care for pregnant women with chronic disease.
  The standard care is given to the participants in the control group. The standard care for pregnant women with chronic disease include five routine visits at a non-specialized midwife and an individually scheduled number of visits with an obstetrician, depending on the type and severity of the chronic Medical disease and possible pregnancy complications.
  The women in the control Group have the same amount of ultrasound examinations as do the women in the intervention Group.
  Women in the control Group can attend auditorium antenatal classes at the hospital.

INTERVENTIONS:
Behavioral: ChroPreg + standard care — * Ongoing update of individual maternity care plan.
  * Extra consultation with the specialized midwife at 20-24 weeks of pregnancy about psychological well-being during pregnancy.
  * Extra consultation with the specialized midwife at 30-33 weeks of pregnancy about individual birth preparation, breastfeeding and post-partum care.
  * Possibility for psychologist consultation.
  * Post-partum: Telephone follow-up by the specialized midwife 1 and 2 weeks after discharge.
  * Postnatal follow-up: 4-6 weeks after delivery: conversation with specialized midwife about the pregnancy and birth.
  Arms: ChroPreg

SUMMARY:
The number of pregnant women affected by chronic diseases such as epilepsy, hypertension and thyroid disease is rising, and in the Danish population 15 % of all pregnant women had a chronic disease in 2016. Chronic disease increase the risk of complications during pregnancy such as preterm birth and caesarian section, while children born of mothers with chronic disease have an increased risk of low birthweight, prematurity and birth effects. Moreover, pregnant women with chronic disease have an increased risk of post-natal depression and report higher rates of anxiety during pregnancy and have described dissatisfaction with the communication with care providers about issues such as breastfeeding, lack of coherence during the course of pregnancy and after delivery.

The purpose of this study is to examine the effect of an increased, interdisciplinary, coordinated and specialized maternity care multimodal intervention for pregnant women with chronic disease on the length of hospitalization (during pregnancy and after delivery). Secondarily, the purpose is to examine the effect of the intervention on psychological well-being and patient satisfaction.

The investigators hypothesis is that the delivery of an increased interdisciplinary, coordinated and specialized intervention targeted pregnant women with pre-existing chronic disease will be beneficial for this group of pregnant women's' length of hospitalization during pregnancy and after delivery due to improved maternity care and improved self-care. Also, the investigators hypothesize that the effect of the intervention will be improved psychological well-being and satisfaction with care during pregnancy and after delivery.

DETAILED DESCRIPTION:
Pregnant women with chronic disease such as epilepsy, sclerosis, hypertension, and thyroid disorders have a significant increased risk of pregnancy complications such as spontaneous abortion, preterm delivery, and caesarian section. Children born by mothers affected by chronic disease have a higher risk of low birthweight, prematurity and birth defects. Moreover women affected by chronic disease have a higher incidence of post-natal depression than women with no history of chronic disease.

Previous studies have found that pregnant some women with chronic disease experienced a lack of continuity in the maternity care: they felt that their different care providers were giving contradictory information on issues such as mode of delivery, breastfeeding and medications. This lack of continuity led to dissatisfaction with care and insecurity with decision-making.

Previous studies that evaluate maternity care interventions, have shown that the elements of the interventions that have a positive effect on pregnancy outcomes such as lowering pregnancy and birth complications, health costs and patient satisfaction are: increased care-coordination, continuity of care providers, specially trained care providers (e.g. nurses and midwives), specialized teams, focus on transitions from e.g. one care setting to another and individualized women-centered care.

However, none of these studies have been targeted pregnant women with chronic disease and how to optimize their course of maternity care. Moreover, systematic reviews point out that studies that examine the effect of the interventions on patient satisfaction, health costs and psychological well-being.

On this background, the purpose of this study is to examine the effect of a midwife-coordinated individualized and specialized maternity care intervention for pregnant women with chronic disease on the length of hospitalization (during pregnancy and after delivery). Secondarily, the purpose is to examine the effect of the intervention on psychological well-being and patient satisfaction.

Patient enrollment The patients will be recruited from the Department of Obstetrics, Rigshospitalet, Denmark from October 2018 to February 2020. Participants will be selected on the basis of 1) the journal information provided from the women's general practitioner and 2) an electronic questionnaire that all pregnant women at Rigshospitalet are sent by e-mail and more than 90% return before 10 weeks of gestation. The information from the questionnaire is routinely transferred to the women's medical journals. Potential participants receive patient information about the study at around week 9-17 of gestation depending on how early the hospital, receive the information about the pregnancy.

The first contact to the patient will be by phone between 12-18 weeks of gestation as a part of the standard care when a midwife from the visitation will call the woman with information about shedueled appointments and programme for high-risk pregnancies at the department. The midwife will ask if information about the study can be sent til the woman and if a research midwife is allowed to follow up on this information with a phone call within a week. If the woman agree, a research midwife will phone the woman within a week and ask if she wants more information about the study and if she wants to participate. If so the woman is given the information and offered the choice between a personal meeting or information over the phone about the study and participation. If the woman agerrs to participate informed concent is obtained, and randomization is performed by a specially designed computer programme.

Data collection. All participants complete an electronic baseline questionnaire after informed consent is obtained and before randomization. All data from the electronically distributed questionnaires are stored in a secured database.

Questionnaire number two (33-37 weeks of gestation) and questionnaire three (two months after delivery) will be sent to the participants by e-mail and the returned questionnaires will be stored in a secured database.

Other data will be obtained from patient records.

Sample size calculation

A total of 258 women will be enrolled in the study. The sample size was determined using unpublished data on 426 pregnant women with chronic diseases hospitalized at Rigshospitalet during pregnancy and in the post-partum period in 2017. The average length of hospital stay (LOS) during pregnancy was 3.9 days; however, due to a right-skewed distribution, log-transformed LOS was used as the outcome for the sample size calculation. Therefore, the effect of the intervention is expressed as a ratio. We expect a reduction of 25% in LOS in the intervention group compared to the control group. This corresponds approximately to a mean reduction of 1 day of hospitalization and to an improvement of log (1-0.25) = -0.29 on the log scale, which we consider a realistic and clinically significant effect size. The SD of number of days in hospital on log scale was 0.80. With a difference of 0.29, SD = 0.80, a power of 0.8 and a significance level of 0.05, an analysis by the two-sample t-test requires 123 women in each group. We expect a maximum of 5% to be lost to follow-up, leading to a total of 129 women needing to be enrolled in each group.

Analysis plan

Analyses are to be performed based on the intention-to-treat principle. The log-transformed number of days in hospital in the two groups will be compared in the primary unadjusted analysis and in a secondary analysis, adjustments will be made for parity and age. Analysis will be performed using the general linear model unless we find a generalized linear model (e.g. Poisson or negative binomial) to fit the distribution of the number of days in hospital. Furthermore, the two groups will be compared with respect to the proportion of women with three or fewer days in hospital. Comparison of secondary and exploratory outcomes will similarly be performed using the general or generalized linear models as appropriate. In case of an uneven allocation of pregnancies with congenital malformations or chromosomal abnormalities to the two groups, analyses will be performed in the sub group of women without pregnancies with congenital malformations or chromosomal abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years and above of age.
* Pregnant women with one or more chronic diseases before pregnancy (e.g. epilepsy, hypertension, lung disease, thyroid disease, multiple sclerosis).
* high-risk pregnancy with planned antenatal care with obstetrician
* Pregnancy with a single fetus.
* Ability to give written informed consent.

Exclusion Criteria:

* Pregnant women below 18 years of age.
* Multiple pregnancies.
* Lack of ability to speak and understand Danish language.
* Substance abuse problems
* Women with diabetes mellitus before pregnancy and women with Heart disease ( these women already receive a special programme at the Deprtment of Obstetrics, Rigshospitalet)
* Chronic psychiatric disease (as only chronic disease)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 262 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization, length of stay (LOS) | 2 weeks post-partum
  The duration of hospitalization will be measured in days (mean and SD)

SECONDARY OUTCOMES:
World Health Organization Five Well-being Index (WHO-5) | 33th-37th week of gestation and 2 months after delivery
  Psychological well-being will be measured by the World Health Organization Five Well-being Index (WHO-5) (mean and SD) or (median and range).
Edinburgh Postnatal Depression Scale (EPDS) | 33th-37th week of gestation and 2 months after delivery
  Symptoms of depression measured by the Edinburgh Postnatal Depression Scale (EPDS) will be defined as cutoff score ≥ 13 and a cutoff score ≥ 10. The scale measures the intensity of common depressive symptoms on a 4-point Likert scale (0-3), where 0 indikates absence of depressive symptoms and 3 indicates the highgest amount of depressive symptoms. The lowest score of the scale is 0 and the highest total score is 30.
Cambridge Worry Scale (CWS) | 33th-37th week of gestation
  The degree of worry during pregnancy measured by the Cambridge Worry Scale (CWS) will be defined as an overall score (mean/SD) or (median/range). The scal consists of a 16 items on a 6-point Likert scale (0-5). The highest total score is 80 indicating the highest level of worry and the lowest score is 0 indicating the lowest level of worry during pregnancy.
Pregnancy & Childbirth Questionnaire (PCQ) | 2 months after delivery
  Patient satisfaction will be measured by the Pregnancy & Childbirth Questionnaire (PCQ) (mean and SD) or (median and range). The scale consists of 25 items on a 5-point Likert scale (0-4). The highest total score is 100 indicating the highest level of satisfaction and the lowest score is 0 indicating the lowest level of satisfaction. The scale can be divided in two subscales. the first subscale measures satisfaction with pregnancy care and education and information and consists of the first 18 items on the total scale. The second subscale measures satisfaction with childbirth and consists of the last 7 items of the total scale.
number of outpatient visits | 2 weeks post-partum
  Outpatient visits will be measured by the number of outpatient visits (mean and SD) or (median and range).
Mode of delivery | 2 weeks post-partum
  Mode of delivery will be measured with respectively spontaneous vaginal delivery, vacuum extraction or caesarian section (n/%)
Onset of labor | 2 weeks post-partum
  Onset of labor will be measures will be measured with respectively spontaneous onset of labor or induced labor (n/%).
Preterm delivery (delivery before 37 full gestational weeks) | 2 weeks post-partum
  Preterm delivery will be measured by yes or no (n/%).
Use of epidural analgesia | 2 weeks post-partum
  Use of epidural analgesia will be measured by yes or no (n/%).
Pregnancy complicated by pre-eclampsia | 2 weeks post-partum
  Pre-eclampsia will be measured by yes or no (n/%l).
Pregnancy complicated by pregnancy-induced hypertension | 2 weeks post-partum
  Pregnancy-induced hypertension will be measured by yes or no (n/%).
Pregnancy complicated with gestational diabetes | 2 weeks post-partum
  Gestational diabetes will be measured by yes or no (n/%).
Birth weight in kilograms | 2 weeks post-partum
  Birth weight will be measured in kilograms (mean and SD).
Newborn's well-being at time of delivery (Apgar-score) | 2 weeks post-partum
  Newborn's well-being at time of delivery will be measured by Apgar-score (yes no to an Apgar-score ≤ 7 at 5 minutes post-partum) (n/%).
  Newborn's well-being at time of delivery will be measured by Apgar-score (yes no to an Apgar-score ≤ 7 at 5 minutes post-partum) (OR and 95 % confidence interval).
Newborn's well-being at time of delivery (pH-value in cord blood) | 2 weeks post-partum
  Newborn's well-being at time of delivery will be measured by the pH-value in the cord blood at time of delivery (mean/SD) or (median and range).
Breastfeeding (2 months after delivery) | 2 months after delivery
  Breastfeeding will be measured by yes/no at 2 months after delivery (n/%).
  Breastfeeding will be measured by yes/no at 2 months after delivery (OR and 95% confidence interval).
  Breastfeeding will be measured by yes/no at 2 months after delivery (OR and 95% confidence interval).
Intention to breastfeed | 33-37 weeks of gestation
  Intention to breastfeed will be measured by yes/no at 33-37 weeks of gestation (N/%).
Intended duration of breastfeeding. | 2 months after delivery
  Intended duration of breastfeeding will be measured in months (mean/SD) or (median and range)
Satisfaction with breastfeeding | 2 months after delivery
  Satisfaction with breastfeeding. Satisfaction with breastfeeding will be measured on a scale from really good to bad (5 categories)(n/%).
Overall satisfaction with maternity care | 2 months after delivery
  Overall satisfaction with maternity care will be measured by percentage of participants in each of the five categories of satisfaction (really good, good, moderate, not so good, poor) (n/%).
Self-evaluated ability to cope with breastfeeding | 2 months after delivery
  Self-evaluated ability to cope with breastfeeding will be measured by percentage of participants in each of the five categories of satisfaction (really good, good, moderate, not so good, poor) (n/%).
Self-evaluated ability to cope with chronic disease | 2 months after delivery
  Self-evaluated ability to cope with chronic disease will be measured by percentage of participants in each of the five categories of satisfaction (really good, good, moderate, not so good, poor) (n/%).
Self-evaluated ability to cope with the mother role | 2 months after delivery
  Self-evaluated ability to cope with the mother role will be measured by percentage of participants in each of the five categories of satisfaction (really good, good, moderate, not so good, poor) (n/%).

OTHER OUTCOMES:
Health related quality af lifeSF-12 | 2 months after delivery
  The SF-12 questionnaire consists of 12 items that measure physical and mental health, divided into eight subscales: physical and social functioning, role limitation due to physical and mental health, bodily pain, general health perceptions (self-rated health), vitality, and mental health. The scores from the subscales can be calculated in two overall scores: Physical Component Summary (PCS) and Mental Component Summary (MCS) with higher scores indicating better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hanne K Hegaard, PhD, Principal Investigator — Department of Obstetrics, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Department of Obstetrics, The Juliane Marie Centre for Women, Children and Reproduction, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Wolff MG, Johansen M, Ersboll AS, Rosthoj S, Brunsgaard A, Midtgaard J, Tabor A, Hegaard HK. Efficacy of a midwife-coordinated, individualized, and specialized maternity care intervention (ChroPreg) in addition to standard care in pregnant women with chronic disease: protocol for a parallel randomized controlled trial. Trials. 2019 May 28;20(1):291. doi: 10.1186/s13063-019-3405-5. PMID 31138296
- Available data/document: Study Protocol — http://doi.org/10.1186/s13063-019-3405-5 — Study Protocol